CLINICAL TRIAL: NCT00986791
Title: Scand-Ankle: A Gold Standard Programme for Alcohol Cessation Intervention in Patients Undergoing Acute Fracture Surgery - A Randomised Clinical Multi-centre Study
Brief Title: Alcohol Cessation Intervention in an Acute Surgical Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Lund University (Other); Hvidovre University Hospital (Other); Esbjerg Hospital - University Hospital of Southern Denmark (Other); National Board of Health, Denmark (Other Government); Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Hanne Tonnesen, Professor, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Scand-Ankle
Record Dates: First submitted 2009-09-29; First posted 2009-09-30 (Estimated); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Acute Fracture Surgery; Alcohol Cessation Intervention; Postoperative Complications; Infection; Ankle Injuries
Keywords: risk reduction
MeSH Terms: conditions — Postoperative Complications; Infections; Ankle Injuries; Risk Reduction Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (No Intervention): Treatment as usual
- GSP-A (Experimental): Gold-Standard-Program for Alcohol cessation intervention (GSP-A): 6-week intensive patient education program with pharmaceutical support
  Interventions: Other: GSP-A

INTERVENTIONS:
Other: GSP-A — 6-week Gold Standard Programme (5 meetings in total) consisting a structured education programme, hotline, thiamine and B-vitamins (300 mg daily), Alcohol Withdrawal Prophylaxis and intervention (Benzodiazepines)and controlled Disulfiram support (200 mg x 2 weekly)
  Other Names: Gold Standard Programme
  Arms: GSP-A

SUMMARY:
Hazardous alcohol intake is an independent risk factor for postoperative complications after major and minor operations, elective and emergency procedures for men and women.

The aim of this study is to evaluate the effect of a 6-week Gold Standard Programme for alcohol cessation intervention in the perioperative period compared to the daily routine guidelines for patients with hazardous alcohol intake undergoing ankle fracture surgery.

ELIGIBILITY:
Inclusion Criteria:

* Drinking 21 or more drinks(one drink containing 12 g ethanol) per week for at least 3 months
* Traumatic ankle fracture requiring internal fixation (osteosynthesis; more than just Kirschner threads or similar minor intervention)
* Informed consent
* Randomisation within 36 hours after entering the orthopaedic department

Exclusion Criteria:

* Major trauma involving other fractures or major lesions,
* Preoperative severe psychiatric disorders (including medicine addiction, severe alcohol dependence [defined as experience of delirium or seizures during abstinence from alcohol], dementia) or other conditions of reduced ability for giving informed consent
* Pathological fractures
* Pregnancy and lactation
* Allergy to benzodiazepines, anaesthesia, pain treatment or disulfiram
* Uncompensated chronic diseases (including fulminate cardiac or liver insufficiency, which are contraindications for disulfiram)
* ASA score 4-5
* Canceled operation
* Withdrawal of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2010-05 (Actual); Primary Completion 2016-01-01 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Postoperative Complications | 6 weeks + 3,6,9 and 12 months
  A composite outcome including postoperative infections, second surgery, dislocated fracture, mal-union and other complications requiring treatment (neurological, pneumonia, thrombosis etc.)

SECONDARY OUTCOMES:
Alcohol Intake | 6 weeks + 3,6,9 and 12 months
  Continuous Alcohol Abstinence: 6 weeks Alcohol Abstinence and low-risk drinking: 3,6,9 and 12 months
Cost-Effectiveness | 6 weeks + 3,6,9 and 12 months
  Cost-Effectiveness regarding postoperative complications and alcohol intake Cost-Utility regarding quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Hanne Tønnesen, Professor, Principal Investigator — WHO-CC, Bispebjerg University Hospital
Locations (3):
- Denmark (3):
  - Hvidovre University Hospital, Hvidovre, Copenhagen
  - Hospital Of South West Denmark, Aabenraa
  - Bispebjerg University Hospital, Copenhagen

REFERENCES:
- [Result] Tonnesen H, Egholm JW, Oppedal K, Lauritzen JB, Madsen BL, Pedersen B. Patient education for alcohol cessation intervention at the time of acute fracture surgery: study protocol for a randomised clinical multi-centre trial on a gold standard programme (Scand-Ankle). BMC Surg. 2015 May 1;15:52. doi: 10.1186/s12893-015-0035-z. PMID 25925742